CLINICAL TRIAL: NCT06532955
Title: Pilot Study on Robotic Assisted Microsurgical Lymphatico-venular Anastomosis
Brief Title: The Robot-LVA Study: Robot-assisted Microsurgical Lymphaticovenous Anastomosis in Breast Cancer-related Lymphedema
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL60199.068.16; METC162053 (Other: Medical Ethical Committee azM/UM)
Record Dates: First submitted 2024-07-15; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Lymphedema; Lymphedema Arm; Lymphedema of Upper Arm; Lymphedema of Upper Limb; Lymphedema; Surgical; Lymphedema, Secondary; Lymphedema of Limb; Lymphedema, Breast Cancer; Lymphedema, Non-Filarial
Keywords: Robot-assisted microsurgery; Microsurgery; Robot; Robotic-assisted; Robot-assisted; Lymphaticovenous anastomosis; Lymphatico-venular anastomosis; LVA
MeSH Terms: conditions — Lymphedema; Neoplasm Metastasis; Breast Cancer Lymphedema; Non-Filarial Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lymphaticovenous anastomosis using Microsure Motion Stabilizer (Experimental): Patients in this group undergo robot-assisted lymphaticovenous anastomosis at one or more locations on the affected arm. The procedure is performed under local anesthesia. Incisions are made at the sites where lymphatic vessels are obstructed, ensuring no harm to the viable part of the lymphatic system. The location(s) are determined prior to surgery using ICG lymphography. LVA(s) are made in the subdermal plane with the aid of a surgical microscope. Generally, 1 to 4 LVAs are made. The LVAs are madeusing a surgical microscope and the operation takes approximately 240 minutes.
  Interventions: Device: Lymphaticovenous anastomosis using Microsure Motion Stabilizer
- Lymphaticovenous anastomosis (Active Comparator): Patients in this group undergo lymphaticovenous anastomosis at one or more locations on the affected arm. The procedure is performed under local anesthesia. Incisions are made at the sites where lymphatic vessels are obstructed, ensuring no harm to the viable part of the lymphatic system. The location(s) are determined prior to surgery using ICG lymphography. LVA(s) are made in the subdermal plane with the aid of a surgical microscope. Generally, 1 to 4 LVAs are made. The LVAs are madeusing a surgical microscope and the operation takes approximately 90 minutes.
  Interventions: Procedure: Lymphaticovenous anastomosis (manual)

INTERVENTIONS:
Device: Lymphaticovenous anastomosis using Microsure Motion Stabilizer — The robot-assisted LVA is performed using the Microsure Motion Stabilizer, a telemanipulation tool that stabilizes a surgeon's movement during open microsurgical operations on extremities, specifically on veins and nerves that are close to the skin.
  The surgeon controls a joystick, which directly copies the surgeon's movements in real-time to an instrument held by the device. The device's software scales down the motions and filters out tremor. Surgical technique and method of treatment are identical to conventional microsurgery. The device is equipped with genuine microsurgical instruments and is compatible with existing surgical microscopes. Instead of holding the instrument directly in hand, which is limited in precision and dexterity, the surgeon operates while the instrument's movements are stabilized. The modular design allows the surgeon to decide what level of manipulation assistance is required during a certain procedure.
  Other Names: LVA; Lympahticovenular anastomosis; Lymphovenous bypass; Lymphatic-venous shunt; Robot-assisted LVA
  Arms: Lymphaticovenous anastomosis using Microsure Motion Stabilizer
Procedure: Lymphaticovenous anastomosis (manual) — Lymphaticovenous anastomosis (LVA) involves connecting a lymphatic vessel to an adjacent vein of similar size, thereby facilitating the outflow of lymphatic fluid in patients suffering from secondary lymphedema
  Other Names: LVA; Lymphaticovenous anastomosis; Lymphovenous bypass; Lymphatic-venous shunt
  Arms: Lymphaticovenous anastomosis

SUMMARY:
This study assesses the performance of robot-assisted microsurgery. Lymphaticovenous anastomosis (LVA) is the most difficult procedure in microsurgery at this moment. The LVA technique is applied to treat for example breast cancer-related lymphedema (BCRL). Therefore, this LVA procedure is compared using a manual expert and the same expert applying robot-assisted LVA.

DETAILED DESCRIPTION:
Microsurgery facilitates procedures such as transplantation of tissue as well as lymphedema treatment. Currently, the plastic surgeon's hands are the limiting factor in microsurgical performance. Robot-assistence increases the movement in precision and might therefore be of great importance for the advancement of microsurgery in the world.

It is a prospective study in Maastricht University Medical Center assessing 60 patients undergoing either robot-assisted or manual lymphaticovenous anastomosis (LVA) tot treat breast cancer-related lymphedema (BCRL). The primary outcome parameter is LVA technique. Secondary outcome measures include duration of surgery, technical errors during & complications peri-operatively, surgeon's satisfaction with the LVA procedure, teh patients' convenience during surgery, arm volume over time and patient's symptoms development over time.

ELIGIBILITY:
Inclusion Criteria:

* Female gender;
* Treated for primary early stage breast cancer;
* Early stage lymphedema of the arm (stage 1 or 2 on ISL classification);
* ELV > 10%;
* Suffering from unilateral disease.

Exclusion Criteria:

* Male gender;
* Stage 3 lymphedema of the arm;
* Receiving current breast cancer treatment;
* Distant breast cancer metastases;
* Current substance abuse;
* History of marcaine or indocyanine green allergy;
* Non-viable lymphatic system as determined by near infrared imaging;
* Previous LVA (<10 years) in the arm with lymphedema.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with breast cancer-related lymphedema
Enrollment: 60 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Efficiency of lymphaticovenous anastomosis (LVA) | Assessed at one moment during, maximally up to 1 year postoperatively
  Efficiency of LVA is measured assessing the quality of the LVA using video recordings of the surgery, which is judged by two independent consultants. The Structured Assessment of Microsurgery Skills (SAMS) measuring method is used to assess the quality of each anastomosis. The SAMS score contains twelve separate items, scored from 1 (bad) to 5 (excellent), grouped into four areas (dexterity, visuo-spatial ability, operative flow and judgement), each subdivided into three technical components.

SECONDARY OUTCOMES:
Duration of the surgery | Assessed once and registered directly after the surgery
  The total duaton of the surgery is from the moment of exploration to find adequate lymph channels and venules to the time to finish the LVA anastomoses during surgery. It is hypothesised that robot assisted surgery will have an equal duration of surgery. The increased precision will compensate the initial extra time for settin up the robotic system
Errors during surgery | Assessed during surgery and registered directly after the surgery on the same day as the surgery
  The SAMS list of peri-operative 'complications' (technical flaws) are judged by the two blinded consultants. The surgeon and research team will also register a list of peri-operative (technical) problems
Perioperative complications | Assessed during surgery and postoperatively, in case any occur
  The surgeon and research team will register a list of peri-operative complications, as well as complications during the full follow-up period.
Surgeon's satisfaction with the procedure | Assessed directly after surgery, on the same day as the surgery
  Is assessed using a ten point Visual Analogue Score. The higher the score, the higher the satisfaction of the surgeon.
Surgeon's learning curve with the procedure in practise | Assessed through study completion, an average of 1 year
  To study the learning curve will be calculated by using a curve fitting method to model learning curves.
Patient's convenience during the surgery | Assessed directly postoperatively,on the same day as the surgery
  Patients' overall convenience during the surgery is assessed using a ten point Visual Analogye Score. The higher the score, the more the patient had experienced during surgery. Moreover, patients are asked to fill in if peculiar matters had occurred which might help to increase the patients overall experience during surgery.
Arm circumference over time | At baseline, 3, 6, and 12 months following LVA
  Arm circumference is assessed by measuring both arms using the Upper Extremity Lymphedema (UEL) index. The arm is measured at 10 and 5 centimeters above and below the elbow, at the elbow, wrist and dorsum of the hand.
Arm volume over time | At baseline, 3, 6, and 12 months following LVA
  Water volumetry assess the arm volume over time
Patient's symptoms over time | At baseline, 3, 6 and 12 months following LVA
  The Lymphoedema Functioning, Disability and Health (Lymph-ICF) questionnaire assesses physical function, mental function, household activities, mobility activities, and life and social activities. This questionnaire is filled in to evaluate the effect of the LVA surgery and is part of the general evaluation of LVA patients. The questionnaire takes approximately five minutes and consists of 29 questions. The score ranges from 0 to 100, with 0 being the highest healthrelated quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Shan Shan Qiu Shao, MSc, PhD, Principal Investigator — Maastricht University Medical Center; Tom van Mulken, MSc, Study Chair — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center+, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The results will be published under an Open Access license, making them accesible to everyone at all times. Requests for sharing individual participant data (IPD) will be evaluated on a case-by-case basis, assessing them for suitable research purposes following the trial's completion.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The data will become available upon request after the completion of the trial and publication of primary manuscripts. Individual participant data will be stored for a period of 15 years.
Access Criteria: Request for data sharing of individual participant data (IPD) will be assessed individuallyn by the principal investigator, considering them for appropriate research purposes after the completion of the trial

REFERENCES:
- [Result] van Mulken TJM, Schols RM, Scharmga AMJ, Winkens B, Cau R, Schoenmakers FBF, Qiu SS, van der Hulst RRWJ; MicroSurgical Robot Research Group. First-in-human robotic supermicrosurgery using a dedicated microsurgical robot for treating breast cancer-related lymphedema: a randomized pilot trial. Nat Commun. 2020 Feb 11;11(1):757. doi: 10.1038/s41467-019-14188-w. PMID 32047155
- [Result] Jonis, Y.M.J., Profar, J. J. A., van Mulken, T. J. M., & Qiu, S. (2023). The MUSA robot and its applicability in lymphatic surgery. Plastic and Aesthetic Research, 10(29), Article A4. https://doi.org/10.20517/2347-9264.2023.06